CLINICAL TRIAL: NCT06414330
Title: Ringer Acetate Based Modified Del Nido Cardioplegia Solution Versus Histidine, Tryptophan and Ketoglutarate Solution Cardioplegia Solution in Cardiac Surgery
Brief Title: Ringer Acetate Based Modified Del Nido Cardioplegia Solution Versus HTK Solution Cardioplegia Solution in Cardiac Surgery
Acronym: HTK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Ahmed Ismail Abdelsabour (Unknown); Ramy Mustafa Abdelgawad Mohamed (Unknown); Ibrahim Mohamed Imbaby (Unknown); Amr Ibrahim Abdelaal (Unknown); Mahmoud Mohamed Atef Sallam (Unknown); Mohamed, Ahmed Abdelhay Mohamed (Unknown)
Responsible Party: Principal Investigator, Ayman Abd El-Khalek Mohammed Glala, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Delnido cardioplegia
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Ischemia
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HTK custidiol (Experimental): will receive HTK (Histidine, Tryptophan and Ketoglutarate solution) consisting of (1000ml distilled water, sodium 15mmol/L, potassium 9mmol/L, magnesium 4mmol/L, calcium 0.015 mmol/L, histidine 129mmol/L, tryptophan 2mmol/L, ketoglutarate 1mmol/L, mannitol 30mmol and pH 7.02 - 1.2). Dose will be 10 - 20 ml/kg and can be repeated once after 120 minutes.
  Interventions: Biological: HTK
- Del Nido (Experimental): will receive modified Del Nido cardioplegia (Ringer acetate 1000ml, mannitol 20% 17 ml, magnesium sulphate 10% 20ml, sodium bicarbonate 8.4% 16ml, potassium chloride 7.5% 13ml and lidocaine 2% 8 ml). Crystalloid to blood ratio will be 80% to 20% respectively. Dose will be 15 - 20 ml/kg in first dose then 8 - 10 ml/kg every 60 minutes
  Interventions: Biological: Ringer acetate based Del Nido cardioplegia

INTERVENTIONS:
Biological: Ringer acetate based Del Nido cardioplegia — All patients will receive hypothermia 29 - 32 ℃ and cardioplegia will be injected between the aortic valve and aortic cross clamp in a pressure not less than 50 mmHg above systolic pressure. After removal of aortic cross clamping, the heart will be monitored for ventricular arrhythmias, early recovery, and postoperative 24 hours serum troponin and new changes in echocardiography.
  Arms: Del Nido
Biological: HTK — Giving HTK instead of Del Nido
  Arms: HTK custidiol

SUMMARY:
Low chloride solutions were proved to be better in resuscitation of emergency cases and decrease the resulting hyperchloremic metabolic acidosis in the last decade. In ringers' acetate solutions, there is acetate, which is metabolized in muscles to produce bicarbonate molecules, so neutralizing the ongoing lactic and hyperchloremic metabolic solutions. Both solutions were proved to be superior to normal saline as a fluid therapy plan in most studies with much less ongoing hyperchloremic metabolic acidosis and inflammatory response. In this protocol, modified Del Nido formula will be involved using ringers' acetate instead of plasmalyte solutions and comparing the effects on myocardial protection versus HTK solutions

DETAILED DESCRIPTION:
First, fulfilling all inclusion criteria and consent acceptance for study are to be confirmed. Preoperative evaluation is done for full laboratory investigations including CBC, coagulation, renal and liver functions, CRP and troponin, full clinical examination for chest and heart, coronary angiography, Echocardiography, carotid doppler and upper and lower venous and arterial doppler are to be done. All patients will be scheduled for on pump CABG surgery. Low dose of midazolam will be given before surgery. Intraoperative monitoring will involve invasive blood pressure, ECG, peripheral pulse oximetry, capnogram.

After induction of anaesthesia and median sternotomy, patients will be randomly allocated into two groups:

Group (D) will receive modified Del Nido cardioplegia (Ringer acetate 1000ml, mannitol 20% 17 ml, magnesium sulphate 10% 20ml, sodium bicarbonate 8.4% 16ml, potassium chloride 7.5% 13ml and lidocaine 2% 8 ml). Crystalloid to blood ratio will be 80% to 20% respectively. Dose will be 15 - 20 ml/kg in first dose then 8 - 10 ml/kg every 60 minutes.

Group (C ) will receive HTK (Histidine, Tryptophan and Ketoglutarate solution) consisting of (1000ml distilled water, sodium 15mmol/L, potassium 9mmol/L, magnesium 4mmol/L, calcium 0.015 mmol/L, histidine 129mmol/L, tryptophan 2mmol/L, ketoglutarate 1mmol/L, mannitol 30mmol and pH 7.02 - 1.2). Dose will be 10 - 20 ml/kg and can be repeated once after 120 minutes.

All patients will receive hypothermia 29 - 32 ℃ and cardioplegia will be injected between the aortic valve and aortic cross clamp in a pressure not less than 50 mmHg above systolic pressure. After removal of aortic cross clamping, the heart will be monitored for ventricular arrhythmias, early recovery, and postoperative 24 hours serum troponin and new changes in echocardiography.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. Any gender
3. Surgery demands cardiopulmonary bypass and cardioplegia.
4. CABG surgeries

Exclusion Criteria:

1. < 18 years old
2. Emergency surgeries
3. Off pump CABG surgeries
4. Taking cardioplegia other than Del Nido or HTK cardioplegia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Any arrhythmia other than sinus rhythm after cross-clamp removal and reperfusion | after aortic declamping and reperfusion of the heart at the end of ischemia time during cardiopulmonary bypass
  Sinus rhythm will be defined by the following criteria: Del Nido cardioplegia vs HTK. Regular rhythm at a rate of between 60 to 100bpm. - Presence of P waves that are followed by a QRS complex at a 1:1 rate. - A PR interval of between 120 and 200ms.

SECONDARY OUTCOMES:
postoperative serum troponin | 24 hour postoperatively
  serum level of troponin in microgram in deciliter
postoperative echocardiography | 24 hour postoperative
  for any new change from preoperative status

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, faculty of medicine, anesthesia and ICU and pain management department, Asyut, Asyut Governorate, Egypt